CLINICAL TRIAL: NCT01985308
Title: A Randomized Double-Blind Sham-Controlled Trial To Evaluate The Treatment Efficacy of Magnetic Resonant Therapy in Autistic Disorder
Brief Title: A Trial To Evaluate The Efficacy of Magnetic Resonant Therapy in Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRT-001
Record Dates: First submitted 2013-11-05; First posted 2013-11-15 (Estimated); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnetic Resonance Therapy (MRT)-Active (Experimental): Magnetic Field, modulated as per EEG analysis, is active for 6 seconds every minute for 30 minutes per day, 5 days per week x 5 weeks.
  Interventions: Device: Magnetic Resonance Therapy (MRT)-Active
- Magnetic Resonance Therapy (MRT)-Sham (Sham Comparator): Magnetic field is not active, but a sham coil is used, for 6 seconds every minute for 30 minutes per day, 5 days per week x 5 weeks.
  Interventions: Device: Magnetic Resonance Therapy (MRT)-Sham

INTERVENTIONS:
Device: Magnetic Resonance Therapy (MRT)-Active
  Arms: Magnetic Resonance Therapy (MRT)-Active
Device: Magnetic Resonance Therapy (MRT)-Sham
  Arms: Magnetic Resonance Therapy (MRT)-Sham

SUMMARY:
The purpose of this study is to show that a magnetic field applied to the front part of the brain of children suffering from Autism Spectrum Disorder(ASD) can improve function and ameliorate symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Autism Spectrum Disorder by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) rendered by the examination and sufficient Childhood Autism Rating Scale 2nd Edition (CARS-2) score to qualify as autism.
* CARS-2 score between 36 and 47 inclusively
* Age between 4 and 12 years (at day of informed consent)
* Child must suffer disrupted sleep patterns defined as a minimum of 3 nights per week of delayed onset of sleep or night-time awakenings. If these are medicated with mild sedatives or melatonin and corrected, the requirement for medication or melatonin will qualify as evidence of a sleep disorder.

Exclusion Criteria:

* Diagnosis of Asperger's Disorder, Pervasive Developmental Disorder Not Otherwise specified
* History of clinically significant traumatic brain injury
* Any condition associated with increased intracranial pressure
* Cerebral Aneurysm
* Down's Syndrome or other chromosomal abnormality
* EEG abnormalities that indicate seizure risk
* Intracranial implant
* Unstable medical condition not otherwise specified
* Clinically significant organic disease unrelated to autism

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Young Kim, MD, Principal Investigator
Locations (2):
- United States (2):
  - Brain Treatment Center, Newport Beach, California
  - Brain Treatment Center of Atlanta, Buford, Georgia

IPD SHARING:
Plan to Share IPD: No
No Identifiable Patient Data (IPD) will be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- MRT-Active: Magnetic Field, modulated as per EEG analysis, is active for 6 seconds every minute for 30 minutes per day, 5 days per week x 5 weeks.
  MRT-Active
- MRT-SHAM: Magnetic field is not active, but a sham coil is used, for 6 seconds every minute for 30 minutes per day, 5 days per week x 5 weeks.
  MRT-SHAM
Period: Overall Study
Arm/Group | MRT-Active | MRT-SHAM
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRT-Active | MRT-SHAM | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.26 (2.53) | 7.64 (2.4) | 7.45 (2.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 10 | 13 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 11 | 19
  Asian/Pacific Islander | 5 | 1 | 6
  Hispanic | 0 | 2 | 2
  African-American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Childhood Autism Rating Scale 2nd Edition (CARS2)
Description: The Childhood Autism Rating Scale is a behavior rating scale that measures the severity of autism symptoms in children. It consists of 15 sub-domains including relating to people, adaptation to change, verbal communication, and visual response. Each sub-domain is rated between 1-4, with the total score ranging from a low of 15 to a high of 60. Scores below 30 indicate that the individual is in the non-autistic range. Scores between 30 and 36.5 indicate mild to moderate autism, and scores from 37 to 60 indicate severe autism. A higher CARS score represents more severe symptoms.
  In the present study, the primary outcome was numerical change in CARS score between baseline and Week 5 (end of the double-blind portion of the study). The comparison of the mean and standard deviation between groups is reported.
  Difference in CARS score between the baseline and week 5 (end of double-blind portion of the study). CARS value at 5 weeks minus CARS value at baseline.
Time Frame: 5 Weeks
Population: Children diagnosed with Autism Spectrum Disorder
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MRT-Active | MRT-SHAM
Number analyzed (Participants) | 14 | 14
units on a scale | -7.68 (4.56) | -1.61 (2.37)
Statistical Analysis 1: Comparison: MRT-Active vs MRT-SHAM; Test type: Superiority; p = 0.0002, t-test, 2 sided

2. Post Hoc Outcome: Child Autism Rating Scale Subdomain Item 7 (Visual Response) - Percent of Subjects Who Improved
Description: Child Autism Rating Scale 2nd Edition (CARS2) consists of 15 Subdomains to rate a child's behavior, characteristics, and abilities against the expected developmental growth of a typical child. This outcome provides the percent of subjects who improved between baseline and Week 10 following all active treatment.
Time Frame: Baseline until after Week 10
Population: Children diagnosed with Autism Spectrum Disorder
Measure: Number; unit: percentage who improved
Groups:
- All Participants Who Completed Week 10: Comprises all study participants who completed Week 10, ensuring that they have received at least 5 weeks of active treatment.
Arm/Group | All Participants Who Completed Week 10
Number analyzed (Participants) | 28
percentage who improved | 71.4

3. Post Hoc Outcome: Child Autism Rating Scale Subdomain Item 11 (Verbal Communication) - Percent of Subjects Who Improved
Description: as for outcome 2
Time Frame: Baseline until after Week 10
Population: Children diagnosed with Autism Spectrum Disorder
Measure: Number; unit: Percentage who improved
Arm/Group | All Participants Who Completed Week 10
Number analyzed (Participants) | 28
Percentage who improved | 66.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 12 weeks.
Arm/Group | MRT-Active | MRT-SHAM
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRT-Active (N=14) | MRT-SHAM (N=14)
Gastrointestinal upset (Gastrointestinal disorders) | 3 (14) | 3 (14)

LIMITATIONS AND CAVEATS:
The small number of patients involved in the study is its primary limitation. One missed aspect was performing a passive cohort EEG analysis of 28 children with autism of the same age, gender and social status who did not undergo MRT treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No